CLINICAL TRIAL: NCT02976116
Title: Fruquintinib in Combination With Gefitinib as First-line Therapy in Patients With Advanced Non-squamous Non-small-cell Lung Cancer Harboring Activating EGFR Mutations : a Single-arm, Multicenter, Phase II Study
Brief Title: A Phase II Study of Fruquintinib in Combination With Gefitinib in Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-013-00CH1
Record Dates: First submitted 2016-11-17; First posted 2016-11-29 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-08

CONDITIONS: NSCLC
Keywords: Fruquintinib; NSCLC; 1st line
MeSH Terms: interventions — HMPL-013; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fruquintinib & Gefitinib (Experimental): Drug: Fruquintinib and Gefitinib
  Interventions: Drug: Fruquintinib; Drug: Gefitinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib will be administered orally once daily from Day 1 to Day 21 per 28-day cycle until disease progression or unacceptable toxicity
  Other Names: HMP-013
Drug: Gefitinib — Gefitinib will be administered orally once daily per 28-day cycle or unacceptable toxicity
  Other Names: Iressa

SUMMARY:
Fruquintinib in combination with Gefitinib as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harboring activating EGFR mutations : a single-arm, multicenter, phase II study

DETAILED DESCRIPTION:
This phase II trial will evaluate the combination of fruquintinib and gefitinib in advanced NSCLC. The endpoint will be to evaluate the efficacy and safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Age between 18 to 75 years old.
* Histologically or cytological documented stage IIIB/IV non-squamous non-small cell lung cancer patients who have never received systematic treatment for the late-stage disease.
* ECOG 0-1
* Patients must have measurable lesions

Exclusion Criteria:

* Prior systematic treatment for the advanced NSCLC
* Absolute neutrophil count (ANC) < 1.5×10^9 /L, or platelet count < 100 ×10^9/L, or hemoglobin < 9 g/dL
* Total bilirubin > 1 ULN; SGOT (AST), SGPT (ALT), > 1.5 ULN; for patient with liver metastasis，AST or ALT > 3 ULN
* Known HIV positive
* Hypersensitivity to either of the investigation drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
tumor objective response rate | Patients will be followed until study completion, an average of 1 year
  Occurrence of completed response or partial response after treatment, assessed by RECIST 1.1
Safety and tolerability | Each patient will be followed for 30 days after the last dose
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Patients will be followed until study completion, an average of 1 year
  The duration from first dose to first documented progression or death from any cause, whichever came first, assessed by RECIST 1.1
Duration control rate (DCR) | Patients will be followed until study completion, an average of 1 year
  Occurrence of completed response, or partial response, or stable disease, assessed by RECIST 1.1
Time to response (TTR) | Patients will be followed until study completion, an average of 1 year
  the period from the date of first dose to the date when the criteria for complete response or partial response was first measured
Duration of response （DoR） | Patients will be followed until study completion, an average of 1 year
  Duration from first documented completed response or partial response to first documented progression or death from any cause, whichever came first

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Yin, Study Director — Hutchison MediPharma Ltd
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - The First Hospital of Zhejiang University, Hangzhou

IPD SHARING:
Plan to Share IPD: No